CLINICAL TRIAL: NCT02211131
Title: A Phase 2, Multicenter, Randomized, Open-label Trial Assessing the Efficacy and Safety of Talimogene Laherparepvec Neoadjuvant Treatment Plus Surgery Versus Surgery Alone for Resectable, Stage IIIB to IVM1a Melanoma
Brief Title: Efficacy and Safety of Talimogene Laherparepvec Neoadjuvant Treatment Plus Surgery Versus Surgery Alone for Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110266; 2014-001146-13 (EudraCT Number)
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Results first posted 2020-05-28 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Completely Resectable Stage IIIB, IIIC, or IVM1a Melanoma
MeSH Terms: interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Other): Surgical resection of melanoma tumor lesion(s)
  Interventions: Procedure: Immediate surgical resection of melanoma lesion(s)
- Talimogene Laherparepvec (Experimental): Talimogene laherparepvec for 6 doses followed by surgical resection of melanoma tumor lesion(s).
  Interventions: Drug: Talimogene Laherparepvec

INTERVENTIONS:
Drug: Talimogene Laherparepvec — Talimogene laherparepvec will be administered by intralesional injection into the injectable cutaneous, subcutaneous, and nodal tumors initially at a dose of 10^6 plaque forming units (PFU)/mL at day 1 of week 1 followed by a dose of 10^8 PFU/mL at day 1 (±3 days) of week 4, 6, 8, 10 and 12 or until all injectable tumors have disappeared, or intolerance of study treatment or in the opinion of the investigator, immediate surgical resection or any other treatment for melanoma is warranted, whichever occurs first.
  Arms: Talimogene Laherparepvec
Procedure: Immediate surgical resection of melanoma lesion(s) — Surgical resection of melanoma tumor lesion(s) will be performed after randomization any time during weeks 1 to 6.
  Arms: Surgery

SUMMARY:
This is a phase 2, multicenter, randomized, open-label study to estimate the efficacy of talimogene laherparepvec as a neoadjuvant treatment followed by surgery compared to surgery alone in subjects with completely resectable stage IIIB, IIIC, or IVM1a melanoma.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, randomized, open-label study to estimate the efficacy of talimogene laherparepvec as a neoadjuvant treatment followed by surgery compared to surgery alone in subjects with completely resectable stage IIIB, IIIC, or IVM1a melanoma.

Arm 1: Talimogene laherparepvec for 6 doses followed by surgical resection of melanoma tumor lesion(s).

Arm 2: Immediate surgical resection of melanoma tumor lesion(s) Following surgery, adjuvant systemic therapy and/or radiotherapy may be administered at the investigator's discretion and per the institutional standard of care.

Subjects will be followed for safety approximately 30 (+15) days after surgery and for disease recurrence, subsequent anticancer therapy, and survival every 3 months (±30 days) for first 3 years after the end of the safety follow-up period and then every 6 months (±30 days) until death, subject withdraws full consent, or up to 5 years after the last subject is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of stage IIIB, IIIC or IVM1a melanoma eligible for complete surgical resection.
* Prior systemic, regional and radiation anticancer therapies for melanoma must have been completed at least 3 months prior to randomization.
* Subject must have measurable disease and must be a candidate for intralesional therapy with at least one injectable cutaneous, subcutaneous, or nodal melanoma lesion (≥ 10 mm in longest diameter) or with multiple injectable lesions that in aggregate have a longest diameter of ≥ 10 mm.
* Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and must have a serum lactate dehydrogenase (LDH) ≤ 1.0 X upper limit of normal and adequate hematologic, hepatic, renal, and coagulation organ function- Other criteria may apply

Exclusion Criteria:

* Subject must not have primary ocular or mucosal melanoma, or history or evidence of melanoma associated with immunodeficiency states (eg, hereditary immune deficiency, organ transplant, or leukemia).
* Subject must not have history or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, or other symptomatic autoimmune disease.
* Subject must not have evidence of clinically significant immunosuppression or active herpetic skin lesions or prior complications of herpes simplex type 1 (HSV-1) infection (eg, herpetic keratitis or encephalitis) and must not require intermittent or chronic systemic treatment with an antiherpetic drug (eg, acyclovir), other than intermittent topical use.
* Subject known to have acute or chronic active hepatitis B, hepatitis C, or human immunodeficiency virus infection will also be excluded.
* Subject must not have been treated previously with talimogene laherparepvec or tumor vaccine.

Other criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (43):
- United States (20):
  - Research Site, Birmingham, Alabama
  - Research Site, Duarte, California
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Santa Monica, California
  - Research Site, Daytona Beach, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Louisville, Kentucky
  - Research Site, Worcester, Massachusetts
  - Research Site, Omaha, Nebraska
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
- Australia (3):
  - Research Site, North Sydney, New South Wales
  - Research Site, Woodville South, South Australia
  - Research Site, Heidelberg, Victoria
- Brazil (3):
  - Research Site, Florianópolis, Santa Catarina
  - Research Site, Barretos, São Paulo
  - Research Site, Rio de Janeiro
- France (5):
  - Research Site, Dijon
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Toulouse
- Greece (2):
  - Research Site, Athens
  - Research Site, Heraklion - Crete
- Poland (3):
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Spain (3):
  - Research Site, Málaga, Andalusia
  - Research Site, Pamplona, Navarre
  - Research Site, Madrid
- Switzerland (2):
  - Research Site, Chur
  - Research Site, Zurich

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Dummer R, Gyorki DE, Hyngstrom J, Berger AC, Conry R, Demidov L, Sharma A, Treichel SA, Radcliffe H, Gorski KS, Anderson A, Chan E, Faries M, Ross MI. Neoadjuvant talimogene laherparepvec plus surgery versus surgery alone for resectable stage IIIB-IVM1a melanoma: a randomized, open-label, phase 2 trial. Nat Med. 2021 Oct;27(10):1789-1796. doi: 10.1038/s41591-021-01510-7. Epub 2021 Oct 4. PMID 34608333
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 35 centers in Australia, Brazil, Europe, Russia, and the United States. Participants were enrolled between 03 February 2015 and 28 April 2022.
Pre-assignment Details: Participants were randomized 1:1 to receive either talimogene laherparepvec for 6 doses followed by surgical resection of melanoma tumor lesions or immediate surgical resection of melanoma tumor lesion(s). Randomization was stratified by disease stage and planned adjuvant therapy.
Groups:
- Surgery: Immediate surgical resection of melanoma lesion(s) any time during Weeks 1 to 6.
- Talimogene Laherparepvec Plus Surgery: Talimogene laherparepvec up to 4.0 mL of 10^6 PFU/mL followed by up to 4.0 mL of 10^8 PFU/mL administered 21 (+5) days after the initial dose. Subsequent doses up to 4.0 mL of 10^8 PFU/mL every 14 (± 3) days until Week 12, all injectable tumors have disappeared, or intolerance of study treatment, whichever occurs first.
  Followed by surgical resection of melanoma lesions(s) anytime during Weeks 13 to 18.
Period: Overall Study
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery
Started | 74 | 76
Completed | 40 | 48
Not Completed | 34 | 28
Not completed — Death | 26 | 16
Not completed — Lost to Follow-up | 4 | 3
Not completed — Decision by Sponsor | 1 | 1
Not completed — Withdrawal by Subject | 3 | 8

BASELINE CHARACTERISTICS:
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (16.1) | 62.6 (12.6) | 60.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 47 | 49 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 69 | 70 | 139
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 73 | 73 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Stratification Factor: Disease Stage [Number; unit: participants] — The clinical participants were staged according to the American Joint Committee of Cancer (AJCC) 7th edition Melanoma Staging System, which combines tumor staging, nodal staging and metastasis to derive an overall stage. The order of prognostication is as follows: stage IIIB (better prognosis) > stage IIIC > stage IV M1a (worse prognosis).
  Randomization was stratified by disease stage and planned adjuvant therapy (adjuvant systemic therapy with or without radiotherapy vs radiotherapy without adjuvant systemic therapy vs none).
  participants
    Stage IIIB Nodal | 14 | 15 | 29
    Stage IIIB In-Transit | 17 | 16 | 33
    Stage IIIC Nodal | 14 | 13 | 27
    Stage IIIC In-Transit With Nodal | 17 | 17 | 34
    Stage IV M1a | 12 | 15 | 27
Stratification Factor: Planned Adjuvant Therapy [Number; unit: participants] — Randomization was stratified by disease stage (IIIB nodal vs IIIB in-transit vs IIIC nodal vs IIIC in-transit with nodal vs IVM1a) and planned adjuvant therapy (adjuvant systemic therapy with (W/) or without (W/O) radiotherapy vs radiotherapy without (W/O) adjuvant systemic therapy vs none).
  participants
    Adjuvant Systemic Therapy W/ or W/O Radiotherapy | 9 | 9 | 18
    Radiotherapy W/O Adjuvant Systemic Therapy | 3 | 3 | 6
    None | 62 | 64 | 126

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-Free Survival (RFS)
Description: Recurrence free survival (RFS) is defined as the time from randomization to the date of event, and is presented as a Kaplan Meier estimate of time to events. The event for RFS is defined as the first of local, regional, or distant recurrence of melanoma or death due to any cause. Participants without a histopathology tumor-free margin (R0) surgical outcome or those who withdrew prior to surgery were considered an event at randomization. Participants without an event were censored at their last evaluable tumor assessment.
Time Frame: 24 months after last participant was randomized (data cutoff date of 30 April 2019)
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 74 | 76
months | 0.0 [NA to NA] — NA=not estimable. There are not enough events to estimate a standard error for the median survival time, confidence intervals (CIs) are not estimable. | 0.0 [0.0 to 6.5]
Statistical Analysis 1: Comparison: Surgery vs Talimogene Laherparepvec Plus Surgery; Test type: Other; p = 0.070, Log Rank — Unstratified log-rank test; Hazard Ratio (HR) = 0.75, 80% CI 2-sided [0.58 to 0.96] — Unstratified Hazard Ratio (T-VEC + Surgery / Surgery)

2. Secondary Outcome: RFS
Description: as for outcome 1
Time Frame: 5 years after the last participant was randomized (last subject last visit occurred 28 April 2022)
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 74 | 76
months | 0.03 [NA to NA] — NA=not estimable. There are not enough events to estimate a standard error for the median survival time, confidence intervals (CIs) are not estimable. | 0.03 [0.03 to 6.54]
Statistical Analysis 1: Comparison: Surgery vs Talimogene Laherparepvec Plus Surgery; Test type: Other; p = 0.092, Log Rank — Unstratified log-rank test; Hazard Ratio (HR) = 0.76, 80% CI 2-sided [0.60 to 0.97] — Unstratified Hazard Ratio (T-VEC + Surgery / Surgery)

3. Secondary Outcome: Kaplan-Meier (K-M) Estimate of RFS Rate at 1 Year, 2 Years, 3 Years, and 5 Years
Description: Kaplan-Meier estimates of the percentage of participants with RFS at 1 year, 2 years, 3 years, and 5 years from randomization. The event for RFS is defined as the first of local, regional, or distant recurrence of melanoma or death due to any cause. Participants without an R0 surgical outcome or those who withdrew prior to surgery are considered an event at randomization. Participants without an event were censored at their last evaluable tumor assessment. Rate is presented as the percentage of participants with RFS at given time point.
Time Frame: 5 years after the last participant was randomized (last subject last visit occurred on 28 April 2022)
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 74 | 76
percentage of participants
  RFS at 1 Year | 21.95 [15.88 to 28.65] | 33.73 [26.82 to 40.76]
  RFS at 2 Years | 16.88 [11.44 to 23.23] | 29.51 [22.91 to 36.40]
  RFS at 3 Years | 16.88 [11.44 to 23.23] | 28.11 [21.62 to 36.94]
  RFS at 5 Years | 15.19 [10.01 to 21.38] | 22.32 [16.39 to 28.84]

4. Secondary Outcome: Histopathology Tumor-Free Margin (R0) Surgical Resection Rate
Description: Histopathology tumor-free margin (R0) surgical resection is defined by pathologist as absence of ink on the tumor for all disease. Rate is presented as the percentage of participants with histopathology tumor-free margin (R0) surgical resection.
Time Frame: 18 weeks after last participant randomized (data cutoff date of 30 April 2019)
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 74 | 76
percentage of participants | 37.8 [30.3 to 45.9] | 42.1 [34.4 to 50.1]
Statistical Analysis 1: Comparison: Surgery vs Talimogene Laherparepvec Plus Surgery; Test type: Other; p = 0.594, Chi-squared — The two-sided p-value is based on the Pearson's Chi-square test; Treatment Difference = 4.3, 80% CI 2-sided [-6.9 to 15.3] — An 80% approximate exact CI for between-arm differences in binary rate is calculated using Wilson's score method with continuity correction

5. Secondary Outcome: Pathological Complete Response (pCR) Rate
Description: Pathological Complete Response (pCR) is defined as no evidence of viable tumor cells on complete pathological evaluation of the surgical specimen per institutional standards of care. Rate is presented as the percentage of participants with pCR.
Time Frame: 18 weeks after last participant randomized (data cutoff date of 30 April 2019)
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 74 | 76
percentage of participants | 2.7 [0.7 to 7.0] | 17.1 [11.6 to 24.0]
Statistical Analysis 1: Comparison: Surgery vs Talimogene Laherparepvec Plus Surgery; Test type: Other; p = 0.003, Chi-squared — The two-sided p-value is based on the Pearson's Chi-square test; Treatment Difference = 14.4, 80% CI 2-sided [7.4 to 21.6] — 80% exact CI for binary rate of each arm is calculated using the Clopper Pearson method

6. Secondary Outcome: Local Recurrence-Free Survival (LRFS)
Description: Local recurrence-free survival (LRFS) is defined as the time from randomization to the earlier date of the first of local disease recurrence or death due to any cause. Participants without an R0 surgical outcome or those who withdrew prior to surgery are considered an event at randomization. Local recurrence is defined as histologically or cytologically confirmed reappearance of melanoma in the area of up to 2 cm from the scar from the surgical excision or at the edge of the skin graft if that was used for closure.
Time Frame: 5 years after the last participant was randomized (last subject last visit occurred on 28 April 2022)
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 74 | 76
months | 0.0 [NA to NA] — NA=not estimable. There are not enough events to estimate a standard error for the median survival time, confidence intervals are not estimable. | 0.0 [0.0 to 7.1]

7. Secondary Outcome: Regional Recurrence-Free Survival (RRFS)
Description: Regional recurrence-free survival (RRFS) is defined as the time from randomization to the date of the first of regional disease recurrence or death due to any cause. Participants without an R0 surgical outcome or those who withdrew prior to surgery are considered an event at randomization. Regional recurrence excludes local recurrence and is defined as histologically, cytologically, or radiographically confirmed reappearance of melanoma in the regional lymph node basin.
Time Frame: 5 years after the last participant was randomized (last subject last visit occurred on 28 April 2022)
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 74 | 76
months | 0.0 [NA to NA] — NA=not estimable. There are not enough events to estimate a standard error for the median survival time, confidence intervals are not estimable. | 0.0 [0.0 to 12.9]

8. Secondary Outcome: Distant Metastases-Free Survival (DMFS)
Description: Distant metastases-free survival (DMFS) is defined as the time from randomization to the date of the first of distant metastases or death due to any cause. Participants without an R0 surgical outcome or those who withdrew prior to surgery are considered an event at randomization. Distant metastases exclude local and regional recurrence and will include distant cutaneous/subcutaneous metastases, distant nodal metastases, or visceral, central nervous system, brain, or bone metastases.
Time Frame: 5 years after the last participant was randomized (last subject last visit occurred on 28 April 2022)
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 74 | 76
months | 0.0 [NA to NA] — NA = not estimable. There are not enough events to estimate a standard error for the median survival time, confidence intervals are not estimable. | 0.0 [0.0 to 6.5]

9. Secondary Outcome: Overall Survival (Kaplan-Meier)
Description: Overall Survival (OS) is defined as the time from randomization to the date of death due to any cause.
Time Frame: 5 years after the last participant was randomized (last subject last visit occurred on 28 April 2022)
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 74 | 76
months | NA [NA to NA] — NA=not estimable. Not enough events occurred to estimate the median and the confidence intervals. | NA [NA to NA] — NA=not estimable. There are not enough events to estimate a standard error for the median survival time, confidence interval is not estimable.

10. Secondary Outcome: Kaplan-Meier Estimate of OS at 1 Year, 2 Years, 3 Years, and 5 Years
Description: Kaplan-Meier estimates of the percentage of participants alive at 1 year, 2 years, 3 years, and 5 years from randomization.
Time Frame: 5 years after the last participant was randomized (last subject last visit occurred on 28 April 2022)
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 74 | 76
percentage of participants
  Year 1 | 85.92 [79.63 to 90.38] | 95.89 [91.58 to 98.02]
  Year 2 | 77.44 [70.29 to 83.08] | 88.94 [83.16 to 92.82]
  Year 3 | 71.59 [64.03 to 77.84] | 83.27 [76.70 to 88.13]
  Year 5 | 62.29 [54.75 to 69.62] | 77.32 [70.12 to 83.00]
Statistical Analysis 1: Comparison: Surgery vs Talimogene Laherparepvec Plus Surgery; Test type: Other; p = 0.050, Log Rank — Unstratified log-rank test; Hazard Ratio (HR) = 0.54, 80% CI 2-sided [0.36 to 0.81] — Unstratified Hazard Ratio (T-VEC + Surgery / Surgery)

11. Secondary Outcome: Best Overall Tumor Response Per Investigator Response Rate (Talimogene Laherparepvec Arm Only)
Description: Response was assessed based on the response of the index lesions and nonindex lesions as described in protocol-defined World Health Organization (WHO) criteria (for complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD]), and presence or absence of new lesions. Best response for a participant is the best overall response observed across all time points. Response rate is reported as the percentage of participants with the best overall response (per investigator) of CR or PR. CR: complete disappearance of all index lesions, including any new measurable tumor lesions which might have appeared. PR: ≥ 50% reduction in the sum of the products of the 2 largest perpendicular diameters of all index lesions and new measurable lesions, if applicable, at the time of assessment as compared to the sum of the products of the perpendicular diameters of all index lesions at baseline.
Time Frame: 18 months after last participant randomized (data cutoff date of 30 April 2019).
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 76
percentage of participants | 13.2 [8.3 to 19.5]

12. Secondary Outcome: Lesion Objective Response Rate: Injected Lesions (Talimogene Laherparepvec Arm Only)
Description: The investigator-assessed tumor response rate for injected lesions, reported as the percentage of evaluable lesions in response. A lesion is in response if the decrease in tumor area is ≥ 50%.
Time Frame: 18 months after last participant randomized (data cutoff date of 30 April 2019).
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Number (80% Confidence Interval); unit: percentage of lesions
Arm/Group | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 76
percentage of lesions | 26.3 [19.7 to 33.9]

13. Secondary Outcome: Lesion Objective Response Rate: Uninjected Lesions (Talimogene Laherparepvec Arm Only)
Description: The investigator-assessed tumor response rate for uninjected lesions, reported as the percentage of evaluable lesions in response. A lesion is in response if the decrease in tumor area is ≥ 50%.
Time Frame: 18 months after last participant randomized (data cutoff date of 30 April 2019).
Population: Intent to Treat Analysis Set: all participants who were randomized to either treatment group.
Measure: Number (80% Confidence Interval); unit: percentage of lesions
Arm/Group | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 76
percentage of lesions | 3.9 [1.5 to 8.6]

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Fatal Adverse Events (AEs), and TEAEs Leading to Discontinuations or Interruptions
Description: Adverse event (AE): any untoward medical occurrence that does not necessarily have a causal relationship with study treatment. SAE: AE meeting at least 1 of the following serious criteria: fatal; life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; congenital anomaly/birth defect; other medically important serious event. Event severity grades: 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening), 5 (death). Treatment begins when the first dose of protocol-required therapies is administered to a participant (Talimogene Laherparepvec Arm) or the participant undergoes surgery (Surgery Arm). Events are reported from first day of study drug or the surgery through 30 days after the last administration of talimogene laherparepvec or 30 days after the surgical resection of melanoma tumor lesion(s), whichever is later.
Time Frame: Adverse Events are reported from first day of study drug or the surgery through 30 days after the last dose of study drug or 30 days after the surgery, whichever is later. Median duration of treatment was 11.14 weeks (range 0.1 to 12.3 weeks).
Population: Safety Analysis Set: all participants who received talimogene laherparepvec (TL) or surgical resection of melanoma tumor lesion(s).
Measure: Count of Participants; unit: Participants
Groups:
- Talimogene Laherparepvec: Pre-Surgery; Talimogene Laherparepvec: Post-Surgery: Talimogene laherparepvec for 6 doses followed by surgical resection of melanoma tumor lesion(s).
  Limited to participants who received at least 1 dose of talimogene laherparepvec and protocol-specified surgery.
Arm/Group | Surgery | Talimogene Laherparepvec: Pre-Surgery | Talimogene Laherparepvec: Post-Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 69 | 57 | 57 | 73
Participants
  All TEAEs | 32 | 53 | 19 | 70
  Grade ≥2 | 19 | 20 | 12 | 38
  Grade ≥3 | 4 | 1 | 7 | 11
  Grade ≥4 | 0 | 0 | 0 | 1
  Serious TEAEs | 2 | 1 | 8 | 13
  Leading to DC of TL | NA — no TL administered | 1 | 0 | 3
  Leading to Interruption of TL | NA — no TL administered | 0 | 0 | 0
  Leading to <4 ml TL Administered | NA — no TL administered | 1 | 1 | 3
  Leading to <4 ml TL Administered: Serious | NA — no TL administered | 1 | 0 | 2
  Leading to <4 ml TL Administered: Nonserious | NA — no TL administered | 0 | 1 | 1
  Fatal Adverse Events | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Talimogene Laherparepvec-Related TEAEs, SAEs, Fatal AEs, and TEAEs Leading to Discontinuations or Interruptions
Description: as for outcome 14
Time Frame: Adverse Events are reported from first day of study drug or the surgery through 30 days after the last administration of talimogene laherparepvec or 30 days after the surgical resection of melanoma tumor lesion(s), whichever is later.
Population: Safety Analysis Set: all participants who received talimogene laherparepvec (TL).
Measure: Count of Participants; unit: Participants
Arm/Group | Talimogene Laherparepvec: Pre-Surgery | Talimogene Laherparepvec: Post-Surgery | Talimogene Laherparepvec Plus Surgery
Number analyzed (Participants) | 57 | 57 | 73
Participants
  All TEAEs | 51 | 0 | 64
  Grade ≥2 | 13 | 0 | 20
  Grade ≥3 | 1 | 0 | 3
  Grade ≥4 | 0 | 0 | 0
  Serious TEAEs | 1 | 0 | 2
  Leading to DC of TL | 1 | 0 | 1
  Leading to Interruption of TL | 0 | 0 | 0
  Leading to <4 ml TL Administered | 1 | 0 | 1
  Leading to <4 ml TL Administered: Serious | 1 | 0 | 1
  Leading to <4 ml TL Administered: Nonserious | 0 | 0 | 0
  Fatal Adverse Events | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events are reported from first day of study drug or the surgery through 30 days after the last dose of study drug or 30 days after the surgery, whichever is later. Median duration of treatment was 11.14 weeks (range 0.1 to 12.3 weeks). All-cause mortality was reported from enrollment through end of follow-up (up to 5 years after randomization).
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all randomized subjects who received talimogene laherparepvec or surgical resection of melanoma tumor lesion(s).
Arm/Group | Surgery | TALIMOGENE LAHERPAREPVEC PLUS SURGERY
All-Cause Mortality (participants affected / at risk) | 26/74 | 16/76
Serious Adverse Events (participants affected / at risk) | 2/69 | 13/73
Other Adverse Events (participants affected / at risk) | 14/69 | 62/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Surgery (N=69) | TALIMOGENE LAHERPAREPVEC PLUS SURGERY (N=73)
Nausea (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound abscess (Infections and infestations) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Device occlusion (Product Issues) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Neck dissection (Surgical and medical procedures) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Surgery (N=69) | TALIMOGENE LAHERPAREPVEC PLUS SURGERY (N=73)
Diarrhoea (Gastrointestinal disorders) | 0 | 8
Nausea (Gastrointestinal disorders) | 1 | 7
Vomiting (Gastrointestinal disorders) | 0 | 7
Chills (General disorders) | 0 | 18
Fatigue (General disorders) | 1 | 20
Influenza like illness (General disorders) | 0 | 26
Injection site erythema (General disorders) | 0 | 4
Injection site pain (General disorders) | 0 | 6
Injection site reaction (General disorders) | 0 | 4
Pain (General disorders) | 6 | 5
Pyrexia (General disorders) | 2 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Dizziness (Nervous system disorders) | 0 | 7
Headache (Nervous system disorders) | 0 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT02211131/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT02211131/SAP_001.pdf